CLINICAL TRIAL: NCT00544258
Title: A Phase I, Pharmacokinetic Study to Evaluate the Extent of Systemic Absorption of PEP005, When Applied as 0.05% PEP005 Topical Gel to a 100 cm2 (5 cm x 20 cm) Contiguous Actinic Keratosis(AK) Treatment Area on the Extensor (Dorsal Aspect) Forearm.
Brief Title: Pharmacokinetic Study to Evaluate the Extent of Systemic Absorption of PEP005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peplin (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-013
Record Dates: First submitted 2007-10-14; First posted 2007-10-16 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2008-05

CONDITIONS: Actinic Keratoses
Keywords: Pharmacokinetic study; Actinic Keratosis; Topical; Dermatology
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Two days consecutive days of application of 0.05% PEP005 Topical Gel to a 100cm2 contiguous AK treatment area of the arm.
  Interventions: Drug: PEP005

INTERVENTIONS:
Drug: PEP005

SUMMARY:
The purpose of this study is to determine the extent of systemic absorption of PEP005 when applied topically for the treatment of actinic keratoses.

DETAILED DESCRIPTION:
Actinic keratoses (AK) is a common skin condition characterized by rough, scaly patches or sores on the top layer of the skin which if left untreated can progress to skin cancer. Current treatments can cause scarring and hypopigmentation, be inconvenient, or require long treatment duration. Non-invasive alternative therapy for treatment of AK lesions is thus being researched.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients at least 18 years of age.
2. A contiguous 100 cm2 treatment area containing at least 5 AK lesions, on the either the right or left extensor (dorsal aspect) forearm.
3. Written informed consent has been obtained.
4. Agreement from the patient to allow photographs of the selected AK treatment area to be taken and used as part of the study package.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the extent of systemic absorption of PEP005 when applied as 0.05% Topical Gel on two consecutive days (Day 1 and Day 2) to a 100 cm2 (5 cm x 20 cm) contiguous AK treatment area on the extensor (dorsal aspect) forearm.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of two consecutive days of application of 0.05% PEP005 Topical Gel, when applied to a 100 cm2 (5 cm x 20 cm) contiguous AK treatment area on the extensor (dorsal aspect) forearm.

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Katsamas, Study Director — Peplin
Locations (1):
- Siller Medical, Silverton Place, 101 Wickham Terrace, Brisbane, Queensland, Australia

REFERENCES:
- See also: Queensland Institute of Medical Research — http://www.qimr.edu.au/